CLINICAL TRIAL: NCT06803316
Title: Optimizing Care Delivery to Support Reengagement in PLWH Returning to HIV Care After Treatment Lapses in Zambia
Acronym: Reengagement
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Washington University School of Medicine (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: REENGAGEMENT (R34); 1R34MH129219-01A1 (NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: HIV Antiretroviral Therapy (ART) Adherence
Keywords: HIV; Antiretroviral Therapy (ART); Retention; Reengagement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 700 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
1.0 Introduction

The scale-up of human immunodeficiency virus (HIV) treatment services has expanded rapidly in Zambia, facilitated by evolution of the HIV response from centralized services to decentralized care and now towards differentiated service delivery models. Nevertheless, optimal effectiveness remains elusive because timely engagement in care to allow uninterrupted access to antiretroviral therapy (ART) and sustained viral suppression remain incomplete1. Ensuring retention in care is especially relevant since greater numbers of HIV-infected patients are also entering a phase of long-term follow-up. After receiving access to HIV care, a high fraction become lost to follow up with some estimates as high as 25-40%2-5, which is defined as the outcome where the patient has missed their appointment by 30 days and has not died or seeking care at a different healthcare facility, or disengaged from care altogether. Research also suggests that LTFU outcomes are driven by a multitude of factors including structural and clinic-based barriers, individual and community-based barriers. A new generation of innovative interventions is needed to overcome these multifaceted barriers to optimization of the engagement of HIV infected patients with the public health systems that have emerged to serve them. Sustained retention is a critical determinant of viral suppression for PLWH, but treatment interruptions put them at high risk for viremia6-16 and mortality17.

Emerging evidence clearly demonstrates that people living with HIV (PLWH) frequently transition in and out of care over time in sub-Saharan Africa6-13,16, and the time of re-engagement in HIV care presents a critical opportunity to break these ongoing cycles of disengagement. Since the presence of specific barriers leads to disengagement from care for some patients, designing strategies targeting these barriers can offer up a natural prospect for ensuring long-term care engagement. It is evident that the strategies required to initiate a patient into care would be markedly different than those to ensure reengagement in care. Even when PLWH return to care after loss to follow-up (LTFU), rates of repeat LTFU in the future are very high18-24. Our preliminary data from Zambia suggests that 30% become LTFU again within 6 months of return, and that 50% of those who are currently LTFU have previously cycled in and out of care5,25. Few interventions have successfully improved return rates among those LTFU9,26,27, but an estimated 50-70% return to care on their own by one year5,28-30. Strategies for intervening at the time of reengagement in care are urgently needed to break these cycles of disengagement in this high-risk population9.

To address these knowledge gaps, we seek to engage key stakeholders in developing a reengagement program to address critical barriers to reengagement and strengthen long-term reengagement in care. This reengagement study will provide important direction for furture interventions and studies to formally test this health-system intervention for patients reengaging in HIV care after LTFU.

1.1 Rationale

Evidence from our groups as well as throughout Africa highlight the critical needs to strengthen programs for reengagement into HIV care. It is well documented that PLWH frequently transition in and out of care over time in sub-Saharan Africa6-13,16 leading to treatment interruptions that can put them at high risk for viremia6-16 and mortality17. Among those who return to care after loss to follow-up (LTFU), rates of repeat LTFU in the future are also very high18-24 with up to 30% becoming LTFU again within 6 months of return. Additionally, among those who are currently LTFU, 50% have previously cycled in and out of care5,25, indicating missed opportunities to intervene. As an estimated 50-70% of those LTFU return to care on their own by one year5,28-30, strategies for intervening at the time of reengagement in care are very promising to help break these cycles of disengagement in this high-risk population9.

1.2 Research Question

What are the most important needs and preferences of patients and providers for a multicomponent reengagement strategy?

2.0 Study Objectives

2.1 Study Specific Aim

To develop a reengagement strategy that meets the needs and preferences of patients and providers in public health HIV settings.

2.2 Scientific Objectives

The study has three main objectives. These include:

1. Assess patient and provider needs and preferences for reengagement strategies using best-worse scaling experiments.
2. Assess patient and provider needs and preferences for reengagement strategies using qualitative methods.
3. Develop an intervention to optimize the experience of reengagement in HIV care using human-centered design.

DETAILED DESCRIPTION:
Purpose of the research: To systematically evaluate the overall patient experience and its effect on retention in care and virologic suppression via multiple novel measurement modalities in public ART clinics in Zambia and make public health HIV treatment more patient centred, manage and enhance perceptions of quality, and strengthen engagement to optimize treatment.

Statement of the problem: Evidence from our previous Betterinfo study (004-06-14) as well as throughout sub-Saharan Africa points to patient experience as a crucial area for improvement. These data offer a simple synthesis and strategy for improvements. That is, when patients perceive encounters with the health system to be high-quality, respectful, accessible, responsive, and effective, engagement is strengthened.

Rationale/Justification for the study: This study will provide important direction for future interventions to implement more patient-centred care in the current public health HIV infrastructure, as it will fill important knowledge gaps regarding clinic-based barriers to care.

Research questions:

1. What are the most important needs and preferences of patients and providers for a multicomponent reengagement strategy?

Main Aim: To develop a reengagement strategy that meets the needs and preferences of patients and providers in public health HIV settings.

Specific objectives: The study has three main objectives. These include:

1. Assess patient and provider needs and preferences for reengagement strategies using best-worse scaling experiments.
2. Assess patient and provider needs and preferences for reengagement strategies using qualitative methods.
3. Develop an intervention to optimize the experience of reengagement in HIV care using human-centered design.

Methodology (design, sampling, data collection methods and tools):

Objective 1: We will conduct best-worse scaling experiments among patients (n=400) and HCWs (n=200) to quantify relative preferences for the contents and implementation attributes for strategies to improve post-return care delivery.

Objective 2: Guided by the Consolidated Framework for Implementation Research44,45 and the Socioecological Model46, we will use qualitative methods to explore how to optimize the experiences of care delivery after returning to HIV care. We will conduct semi-structured interviews with PLWH who reengaged in the past 6 months and did (n=15) and did not (n=15) remain in care as well as focus group discussions with HCWs (i.e., physicians, nurses, clinic leadership; 6 FGDs, n=8-10 each)

Objective 3: Using principles from human-centered design47,48 and intervention mapping49, we will synthesize findings from Aim 1 and co-develop a multicomponent reengagement coordination implementation strategy focused on:

1. improving the patient experience of reengagement,
2. optimizing ART re-initiation and viral load monitoring post-return, and
3. offering services tailored to initial LTFU reasons to support sustained engagement.

We employ an iterative human-centered process involving key stakeholders (reengaged PLWH, HCWs, clinic leadership, Ministry of Health) to co-design the key components (e.g., practice facilitation and audit-feedback for providers, tailored services for patients) and develop a locally appropriate and acceptable intervention prototype.

Data management issues (data management plan, analysis and storage):

Objective 1: We will summarize routine survey responses using frequency and proportions. We will evaluate the BWS exercise using count analysis and BWS scores for individuals (difference in number of times item scored best and worst/number of times item appears) and, aggregate score for the population (mean population score f rescaled to 100, presented as forest plots). We will use standard statistical techniques to explore preference heterogeneity and we will perform subgroups analyses across characteristics including reason for initial LTFU (i.e., structural, clinic-based, psychosocial), sex, age, and HCW cadre. Data will be kept in a secure and locked file until the interviews are transcribed and the transcription is finalised, after which the recordings and notes will be destroyed. Data will be kept in a password-protected computer file that will only be accessible to members of the research team for data analysis. Once data are linked to SmartCare records using ART numbers, identifying information will be removed in order to maintain confidentiality.

Objective 2: Recordings will be transcribed by trained CIDRZ RAs, and if necessary, translated into English with subsequent back translation or a second-party review of sections of the translation. With the transcribed audio-recording data, we will code and computerize for analysis. The audio recordings, data collection tools and memos will be kept in a secure and locked file until the interviews are transcribed and the transcription is finalised, after which the recordings and notes will be destroyed. Identifying information will be removed during transcription in order to maintain confidentiality. Transcriptions will be kept in a password-protected computer file that will only be accessible to members of the research team for data analysis. Investigators will use thematic content analysis across all data to analyse the data using qualitative software (e.g. Dedoose or NVivo). Qualitative data analysis consists of searching for patterns in data and conceptualizing ideas that help explain the presence of those patterns. For patient interviews, we will also employ a narrative analysis where we read each interview as a whole, without regard to individual codes, to create a more global understanding of the "point of the story".

Objective 3: Implementation of HCD generally follows an iterative framework of inquiry, problem-solving and co-design. Diverse methods are employed in each of these phases including system/stakeholder mapping, compiling secondary data, user journey maps/personas, cognitive sorting and ranking, and iterative prototyping5,118-120. We will collect detailed meeting minutes, visual outputs created from participatory activities, written reflections from participants, and take careful notes during the design team meetings and workshops. We will qualitatively analyze data gathered during the HCD co-creation activities using affinity mapping and rapid thematic analysis. This will occur in between co-creation workshops to identify design opportunities to discuss in future workshops and also after the close of the final workshop.

Participants to be recruited and inclusion criteria: This study will be conducted in Lusaka province at four Ministry of Health-operated facilities that are supported by the Centre for Infectious Disease Research in Zambia (CIDRZ). All participants must give consent to participate. Additional inclusion criteria, sampling and sample size are as follows:

Objective 1 PLHW reengaging in HIV care: We will enrol up to 400 PLWH (age≥18 years) who are reengaging in care from four health care facilities supported by CIDRZ in Lusaka. Reengaging in care will be defined as returning to care after being considered LTFU, which is defined as being greater than 60 days late to their last appointment per Zambian HIV guidelines105. We will include PLWH returning to their original clinic or as a transfer from a different facility. We will recruit participants on the day of return to care using similar recruitment procedures as Objective 1. Eligible participants will be identified by clinical staff during their routine clinic visit, and trained CIDRZ research assistants (RAs) will then recruit and enroll them in a private area as they wait for their clinical consultation or drug pick-up. We have used this approach to successfully recruit over 300 returning patients to date as part of an ongoing study (BMFG OPP1166485).

Healthcare Workers: We will enrol up to 200 health care workers who participate in the care of PLWH across these four health care facilities. This includes clinic leadership (i.e., in-charge), medical officers, clinical officers, nurses, lay health care workers, and pharmacists. We use convenience sampling to identify HCW for surveys using procedures that have been well-established by our study team82,95 in Zambia to successfully recruit HCWs. We will first engage with clinic leadership to identify appropriate times for recruitment and survey administration.

Objective 2 Patient Semi-Structured Interviews: We will recruit PLWH (age≥18 years) who reengaged in care within the past 6 months at four health care facilities supported by CIDRZ in Lusaka and subsequently did (n=15) and did not (n=15) remain in care. We will recruit individuals amongst our survey cohort who agreed to be contacted in the future for qualitative interviews. Reengaging in care will be defined as returning to care after being considered LTFU, which is defined as being greater than 60 days late to their last appointment per Zambian HIV guidelines105. We will include PLWH returning to their original clinic or as a transfer from a different facility. We will use purposive and maximum variation sampling of participants106-108 to ensure participants represent a range of perspectives (i.e., we will recruit participants based on patient characteristics such as gender and age to ensure a range of perspectives as well as barriers to care identified during surveys in Objective 1).

Eligible participants who remained in care will be identified by clinical staff during their routine clinic visit, and trained CIDRZ research assistants (RAs) will then recruit and enroll them in a private area. Those who become LTFU within 6-months of return will be identified in the EHR, through clinic logs, and through routine tracing procedures already in place. These individuals will be contacted via phone and recruited; if they agree to participate, they will then be interviewed in-person in mutually agreed private location. Our research team and CIDRZ has previously used these procedures to recruit LTFU participants for in-depth interviews58,68.

Healthcare workers: The target population for this objective are all health care workers delivery HIV care at our study facilities. This includes clinic leadership (i.e., in-charge), medical officers, clinical officers, nurses, lay health care workers, and pharmacists. We use convenience sampling to identify HCW for focus groups discussions among HCWs (i.e., clinicians, nurses, lay HCWs, pharmacists, clinic leadership) at four facilities. We will use procedures that have been well-established by our study team82,95 in Zambia to successfully recruit HCWs. We will first engage with clinic leadership to identify appropriate times for recruitment and interviews. We will conduct 6 FGDs (N=8-10 each), which will be organized by HCW cadre to ensure that there is open discussion with minimal concern for power hierarchies.

Objective 3 We will recruit reengaged patients (beneficiaries) and HCWs (implementers). Informed by Aim 1 findings, we will also use stakeholder mapping to identify key groups who may influence reengagement behaviors and outcomes among PLWH and HCWs and purposefully recruit from these groups from the four facilities in Aim 1. A priori, we expect to engage with patients who have reengaged in care (n=5-10), health care workers (n=5-10) (as beneficiaries and implementers, respectively, of the interventions) and clinic leadership (n=5) and Ministry of Health administrators (n=1-2) as influencers. Our team has experience recruiting and engaging these multilevel stakeholders in HCD workshops82. Recruitment will be similar to procedures outlined in previous objectives. Participants will be given K100 for travel reimbursement.

Ethical considerations: We submit the proposed protocol, the informed consent documents, data collection tools and any subsequent modifications for review and approval. Also, the Washington University School of Medicine (WUSM) Institutional Review Board (IRB) will provide ethical reviews and regulatory oversight through a reliance agreement with the other collaborating US institutions. We request an expedited review. We will obtain written informed consent from participants agreeing to participate in the following study activities:

* Patient Surveys and In-depth Interviews with patients.
* Health care worker surveys and Focus group discussions

Permission will be sought from national, provincial, district and facility Ministry of Health authorities to conduct the study in public health facilities. The study will follow standard Ministry of Health guidelines to engage with staff, patients and patient records. We will also ensure that all staff involved with study data are trained in Good Clinical Practice and Human Subjects Protection.

Timelines: The study proposes to implement the study intervention over a course of 18 months. Detailed timeline with activities are outlined in the proposed protocol.

Plans to disseminate research findings:

In-order to maximise the benefit of the study findings without delay, the study findings will be shared with key stakeholders such as Ministry of Health and community leaders. Study findings will be disseminated at national, international meetings, conferences and in scientific journals. Permission will be sought from National Health Research Authority prior to any publications or any form of dissemination being made.

POSSIBLE BENEFITS TO PARTICIPANTS:

No direct benefits to participants are expected. Participants may benefit in that the aim provides a direct outlet for their input to be translated into intervention design and future policy decisions. Participants may benefit from improvements in quality of care provided and increased understanding from health care workers resulting from this work. Those disengaged from care may benefit from tracing and follow up by trained counsellors and may decide to re-engage in care. Participants will also receive a small reimbursement (approximately K 100) for their transport and time spent to participate in semi-structured interviews or FGDs. Health care workers and facilities may benefit from understanding patient expectations and from learning how data can be used to interpret and improve clinic practices. Patients may also benefit from the knowledge that their perspectives are valued for improving care delivery. The Zambian Ministry of Health will benefit from the coaching provided by the research team, which may serve to improve the working environment for health care workers and care delivered to patients. The HCD process will result in developing a reengagement strategy that can improve the care of people living with HIV.

POSSIBLE RISKS TO PARTICIPANTS:

All interviews and discussion have the potential to make participants embarrassed, worried, anxious, or uncomfortable when reporting on their interactions. Participants may feel uncomfortable answering questions or discussing their HIV treatment history with the research team during semi-structured interviews or when completed surveys. The research staff will be trained to be sensitive to these areas, for example, such as discussing challenges with HIV care, livelihoods, or family. HCWs may similarly experience discomfort discussing or answering surveys pertinent to their own skills or work preferences. Some participants who are currently lost from care may be contacted via telephone to participate in interviews. This contact may have a small possible risk of involuntary disclosure of HIV status. We will attempt to minimize this by training all follow up staff to be discrete and professional, ensuring that patient confidentiality is maintained at all times and identities are verified prior to providing additional information.

During FGDs, colleagues may also be present and HCWs may fear reprisal if confidentiality is breached. FGDs will be organized by HCW cadre to be sensitive of power dynamics and ensure comfort in openly discussing pertinent topics.

Participants in HCD workshops may also feel uncomfortable answering questions and participating in discussions regarding the challenges about receiving and/or delivering HIV care. Patients may fear negative attitudes from HCWs and HCWs may worry about retribution from their superiors. Workshop composition will be attentive to power dynamics, ensuring participants are engaged on days of the workshop or through sub-groups such that they are free to share their opinions and act as co-designers (e.g., patients or HCWs feel free to share thoughts in presence of health care administrators).

Details of how these risks will be minimised are outlined in the protocol.

POSSIBLE BENEFITS TO THE COMMUNITY:

The potential benefits to society may be an increased understanding of how the process of reengagement can be improved to facilitate ongoing sustained engagement in care and overall HIV outcomes and the needs and preferences of key stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be over 18 years of age.
* Should be LTFU for greater than 30 days or
* Should not have had ART drugs for greater than 30 days;
* Pregnant women who meet inclusion criteria
* Illiterate participants willing to provide informed consent in Nyanja or Bemba provided there is a witness.

Exclusion Criteria:

* Participant is too sick i.e., failing to talk, general discomfort and emergency cases).
* Participant is unable to provide written informed consent in English, Nyanja or Bemba.
* Participant who is drunk or mentally ill.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient Semi-Structured Interviews: We will recruit PLWH (age≥18 years) who reengaged in care within the past 6 months at four health care facilities supported by CIDRZ in Lusaka and subsequently did (n=15) and did not (n=15) remain in care. We will recruit individuals amongst our survey cohort who agreed to be contacted in the future for qualitative interviews. Reengaging in care will be defined as returning to care after being considered LTFU, which is defined as being greater than 30 days late to their last appointment per Zambian HIV guidelines105 and or not having ART drugs for greater than 30 days.
  Healthcare workers: The target population for this objective are all health care workers involved in delivery HIV care at our study facilities. This includes clinic leadership (i.e., in-charge), medical officers, clinical officers, nurses, lay health care workers, and pharmacists. We use convenience sampling to identify HCW for in-depth interviews (IDIs) (i.e., clinicians, nurses,
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Retention | 2022 to 2025
  Those who are less than 30 days late to their scheduled appointments and consistently taking their medication

CONTACTS AND LOCATIONS:
Overall Officials: Izukanji Sikazwe, Medical Officer, Principal Investigator — Centre for Infectious Disease Research in Zambia (CIDRZ)
Locations (1):
- Centre for Infectious Disease Research in Zambia (CIDRZ), Lusaka, Lusaka Province, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Data will be kept in a secure and locked file until the interviews are transcribed and the transcription is finalised, after which the recordings and notes will be destroyed. Data will be kept in a password-protected computer file that will only be accessible to members of the research team for data analysis. Once data are linked to SmartCare records using ART numbers, identifying information will be removed in order to maintain confidentiality. Similarly, transcriptions will be kept in a password-protected computer file that will only be accessible to members of the research team for data analysis.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 2022 - 2025